CLINICAL TRIAL: NCT05341037
Title: A Novel Biomarker for the Prediction of Early Comorbidity in Cardiac Surgery: Red Cell Distribution With to Lymphocyte Ratio
Brief Title: Red Cell Distribution With to Lymphocyte Ratio in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balcı, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: MH2.7
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Surgery
Keywords: red cell distribution width; lymphocyte; postoperative complications; cardiac surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative complications +: Patients who have postoperative complications during hospital stay after cardiac surgery
- Postoperative complications -: Patients who have not postoperative complications during hospital stay after cardiac surgery

SUMMARY:
It is aimed to investigate whether red cell distribution with (RDW) to lymphocyte ratio (RLR) can predict early comorbidity among cardiac surgery patients.

DETAILED DESCRIPTION:
There are important developments in the field of cardiac surgery due to advances in medical treatments, surgical techniques, intraoperative anesthesia management, and postoperative intensive care. On the other hand, the proportion of high-risk patients has increased due to the increasing number of elderly patients with comorbidities presenting for cardiac surgery. It is important to analyze outcomes such as postoperative morbidity and mortality, due to concerns about the quality of life of patients after cardiac operations, the recommendations of current ERAS protocols, and the shortening of intensive care unit length of stay. Complications such as cardiac, pulmonary, renal, and neurological disorders, infections such as pneumonia or sepsis, and prolonged stay in the intensive care unit and hospital are indicators of not only the quality of care but also the quality of life after cardiac surgery. Therefore, it is important to determine the perioperative risk factors that cause postoperative morbidity. Various outcome prediction models are used for cardiac surgery, such as the Cardiac Anesthesia Risk Assessment score, Tuman score, Tu score, and the European System for Cardiac Operative Risk Assessment score, which uses preoperative factors to predict the postoperative outcomes. It is known that intraoperative factors such as CPB duration, aortic cross-clamp time, surgical technique, and serum lactate levels are associated with postoperative morbidity. Recent studies suggest that inflammatory and immune imbalance may play an important role in postoperative complications. Studies point to new parameters derived from preoperative complete blood count as potential biomarkers of inflammation and oxidative stress. Many markers such as Neutrophil/Lymphocyte ratio, Mean platelet volume (MPV) or RDW alone have been studied in cardiac surgery. The ratio of red cell distribution width (RDW) to lymphocyte (L) has been popular in recent years as an indicator of poor prognosis, especially in oncological patients. However, this marker has not yet been evaluated in terms of morbidity or mortality in cardiac surgery patients.

The main purpose of this study; To investigate the RDW/L ratio as an early morbidity marker in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing open-heart surgery with cardiopulmonary bypass

Exclusion Criteria:

* Re-operations
* Emergency operations
* Patients with preoperative renal failure
* Patients with preoperative hematological problems
* Patients with preoperative infection
* Patients with preoperative immunological disease
* Patients using preoperative steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone open-heart surgery with cardiopulmonary bypass in our hospital within the last year will be evaluated retrospectively.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
red cell distribution width (RDW) | preoperative period ( 24 hours before surgery)
  preoperative measurement of complete blood count. RDW is calculated by dividing the standard deviation of the mean cell size by the MCV of the red cells and multiplying by 100 to convert to a percentage.
lymphocyte count | preoperative period ( 24 hours before surgery)
  preoperative measurement of complete blood count.
Complications | postoperative periods, up to 7 days
  postoperative complications such as pulmonary, neurologic, cardiac, infectious.

CONTACTS AND LOCATIONS:
Overall Officials: ZELİHA A DEMİR, Professor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Aydinli B, Demir A, Guclu CY, Bolukbasi D, Unal EU, Koculu R, Selcuk G. Hematological predictors and clinical outcomes in cardiac surgery. J Anesth. 2016 Oct;30(5):770-8. doi: 10.1007/s00540-016-2197-y. Epub 2016 Jun 9. PMID 27282623
- [Result] Unal EU, Ozen A, Kocabeyoglu S, Durukan AB, Tak S, Songur M, Kervan U, Birincioglu CL. Mean platelet volume may predict early clinical outcome after coronary artery bypass grafting. J Cardiothorac Surg. 2013 Apr 16;8:91. doi: 10.1186/1749-8090-8-91. PMID 23590976
- [Result] Huang J, Zhao Y, Liao L, Liu S, Lu S, Wu C, Wei C, Xu S, Zhong H, Liu J, Guo Y, Zhang S, Gao F, Tang W. Evaluation of Red Cell Distribution Width to Lymphocyte Ratio as Potential Biomarker for Detection of Colorectal Cancer. Biomed Res Int. 2019 Jul 31;2019:9852782. doi: 10.1155/2019/9852782. eCollection 2019. PMID 31467924
- [Result] Ma C, Liu Q, Li C, Cheng J, Liu D, Yang Z, Yan H, Wu B, Wu Y, Zhao J. Novel Blood Indicators of Progression and Prognosis in Renal Cell Carcinoma: Red Cell Distribution Width-to-Lymphocyte Ratio and Albumin-to-Fibrinogen Ratio. J Oncol. 2020 Nov 25;2020:2895150. doi: 10.1155/2020/2895150. eCollection 2020. PMID 33299415